CLINICAL TRIAL: NCT07364591
Title: Immediate Effect of Kinesiotaping With Rounded Shoulder Posture in University Students: A Randomized Sham-Controlled Study
Brief Title: Immediate Effect of Kinesiotaping With Rounded Shoulder Posture in University Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Zehra KORKUT, Dr., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000-0001-9243-0937
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Rounded Shoulder Posture; Kinesio Taping
Keywords: Posture; Kinesiotaping; students

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping Group (Experimental)
  Interventions: Other: Kinesiotaping
- Sham Group (Sham Comparator)
  Interventions: Other: Kinesiotaping(no tension)

INTERVENTIONS:
Other: Kinesiotaping — Elastic kinesiology tape will be applied by a licensed physiotherapist with experience in taping. With the participant standing in scapular retraction and neutral posture, a Y- or I-strip is placed from the anterior aspect of the acromion toward the spinous process of T10, with 30-40% stretch over the mid-portion and 0% tension on anchors. A second overlay strip will be applied along the same path with 30-40% stretch to augment the mechanical cue. Skin will be cleaned and dried; hair trimmed if needed. Tape will be rubbed to activate adhesive. Total application time ≈3-5 minutes. Tape remains in place during immediate (≤3 minutes) and short-term (~30 minutes) assessments and is then removed. Adverse skin reactions will be monitored; tape will be removed immediately if irritation occurs.
  Arms: Kinesiotaping Group
Other: Kinesiotaping(no tension) — The sham application is performed in the same area and configuration as the experimental arm; however, the strip is applied completely without tension (0%) along its length and does not provide a therapeutic mechanical cue. To maintain blinding, a second strip is applied along the same path with 0% tension and approximately 50% overlap. Skin preparation and application-removal procedures are identical to the experimental condition. The tape remains in place during the immediate (≤3 minutes) and short-term (~30 minutes) assessments and is then removed.
  Arms: Sham Group

SUMMARY:
Posture is maintained through the interaction of the musculoskeletal system, visual input, vestibular function, and proprioception to provide optimal balance with minimal energy expenditure. Various factors, including prolonged static sitting, unsuitable work environments, prolonged screen use, and low physical activity levels, may contribute to postural misalignment, particularly in student populations. Rounded shoulder posture is commonly associated with muscle imbalance, altered scapular alignment, pain in the neck and shoulder region, reduced range of motion, and functional limitations.

Kinesio taping is a physiotherapy intervention commonly used in orthopedic and musculoskeletal rehabilitation. Proposed effects include facilitation of proper muscular and fascial alignment, enhancement of proprioceptive feedback, and potential improvement in posture and movement quality. However, evidence regarding the immediate effects of kinesio taping on posture-related outcomes in individuals with rounded shoulder posture remains limited.

The purpose of this study is to evaluate the immediate effects of kinesio taping on posture, shoulder range of motion, and proprioception in students with rounded shoulder posture.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-30 years of age
* Having an acromial distance ≥ 2.6 cm measured in the supine position with shoulders in a neutral position

Exclusion Criteria:

* Having a surgical or pathological/neurological condition in the shoulder or spine region (rotator cuff repair, subacromial impingement syndrome, acute tendinitis, cervical disc herniation, scoliosis, fibromyalgia, etc.)
* Having a neurological/systemic disease that may cause sensory problems
* Having an allergic reaction to the use of the tape
* Having a skin lesion, open wound, or skin infection at the taping site
* Using medication within the last 24-48 hours
* Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
posture assessment | Baseline (pre-taping), immediately after application, and 30 minutes post-application.
  PostureScreen Mobile is a valid and reliable mobile application that provides clinical-level postural assessment and analysis. The application uses photographs captured with a mobile device camera from anterior, lateral, and posterior views to evaluate body alignment, asymmetries, and postural deviations. Through visual analysis, the application performs angular and linear measurements to support objective postural evaluation.
  Planned measurement parameters include head translation (cm), head tilt angle, shoulder translation (cm), shoulder tilt angle, rib cage translation (cm), rib cage tilt angle, pelvic translation (cm), pelvic tilt angle, craniovertebral angle, kyphosis angle, and pelvic tilt. To ensure measurement consistency, the mobile device camera position will be standardized at a fixed distance and height for all participants. To enhance visibility and measurement accuracy, participants will be assessed barefoot and wearing only underwear during photographic capture.

SECONDARY OUTCOMES:
Assessment of Joint Range of Motion | Measured at baseline, immediately after taping (≤3 minutes), and 30 minutes post-taping; primary comparison is change from baseline
  Shoulder range of motion will be assessed using the Goniometer Pro smartphone application, which provides valid and reliable angular measurements. Shoulder flexion and extension, abduction and adduction, and internal and external rotation will be evaluated.
  For each measurement, the smartphone will be securely fixed to the segment being assessed and calibrated to zero in the neutral position. During shoulder flexion and abduction measurements, the device will be positioned on the lateral surface of the humerus. For internal and external rotation measurements, the device will be placed on the dorsal surface of the forearm (ulna) with the shoulder positioned at 90 degrees of abduction.
  Participants will be aligned in standardized test positions, and compensatory movements, including scapular elevation and lumbar extension, will be manually restricted. The limb will be moved to the end range of the target motion, and the angular value will be recorded. Each measurement will be repeated
Pressure pain threshold | Measured at baseline, immediately after taping (≤3 minutes), and 30 minutes post-taping; primary comparison is change from baseline
  Pressure pain threshold measurements will be performed bilaterally on the dominant and nondominant sides using a digital algometer (JTECH Medical, Commander Echo). Due to increased activity and sensitivity of the upper trapezius muscles in individuals with rounded shoulder posture, assessments will be conducted on the upper trapezius muscle.
  During digital algometry, pressure will be applied to the measurement site at a constant rate of approximately 1 kg/s. The pressure value at which pain is first perceived will be recorded. Three consecutive measurements will be obtained, and the mean value will be used for analysis.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barker V. Postura, posizione, movimento. Roma: Edizioni Mediterranee; 1998. ISBN: 9788827212165. Kendall FP, McCreary EK, Provance PG. Muscles: Testing and Function with Posture and Pain. 5th ed. (Port.) São Paulo: Manole; 2007. Carini F, Mazzola M, Fici C, Palmeri S, Messina M, Damiani P, et al. Posture and posturology, anatomical and physiological profiles: overview and current state of art. Acta Biomed. 2017;88(1):11-16. doi:10.23750/abm.v88i1.5309. PMID: 28467328; PMCID: PMC6166197. Zhang C, Zhang J, Yang G. Association between internet addiction and the risk of upper cross syndrome in Chinese college students: A cross-sectional study. Medicine (Baltimore). 2023;102(30):e34273. doi:10.1097/MD.0000000000034273. PMID: 37505162; PMCID: PMC10378816. Silva AG, Punt TD, Sharples P, Vilas-Boas JP, Johnson MI. Head posture and neck pain of chronic nontraumatic origin: a comparison between patients and pain-free persons. Arch Phys Med Rehabil. 2009;90(4):669-674. doi:10.1016/j.apmr.2008.10.018. PMID: 19345785. Kim EK, Kim JS. Correlation between rounded shoulder posture, neck disability indices, and degree of forward head posture. J Phys Ther Sci. 2016;28(10):2929-2932. doi:10.1589/jpts.28.2929. PMID: 27821964; PMCID: PMC5088155. Kase K, Wallis J, Kase J. Clinical Therapeutic Applications of the Kinesio Taping Method. Tokyo: Ken Ikai Co.; 2003. Cho HY, Kim EH, Kim J, Yoon YW. Kinesio taping improves pain, range of motion, and proprioception in older patients with knee osteoarthritis: a randomized controlled trial. Am J Phys Med Rehabil. 2015;94(3):192-200. doi:10.1097/PHM.0000000000000148. PMID: 25706053. Toprak Celenay S, Ozkan T, Unluer NO. Short-term effects of trunk kinesio taping on trunk muscle endurance and postural stability in healthy young adults: A randomized controlled trial. Fizyoterapi Rehabilitasyon. 2019;30(2):89-96. doi:10.21653/tfrd.437491.